CLINICAL TRIAL: NCT02044341
Title: A Phase 3, Multicenter, Placebo-controlled, Double-blind, Randomized Study to Compare the Efficacy and Safety of AR01 Otic Solution to a Placebo Solution for Relief of Pain in Acute Otitis Media Subjects Aged 2 Months to 19 Years
Brief Title: Phase 3 Study to Compare the Efficacy and Safety of AR01 to a Placebo Solution for Relief of Pain in Acute Otitis Media
Acronym: AR01006
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Arbor Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AR01.006
Record Dates: First submitted 2014-01-22; First posted 2014-01-24 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-03

CONDITIONS: Acute Otitis Media
Keywords: Acute Otitis Media; Pain; Ear Pain; Ear Ache; Ear infection; middle ear infection
MeSH Terms: conditions — Otitis Media; Pain; Earache; Otitis | interventions — Benzocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AR01 - Topical Otic Solution (Active Comparator): Topical ear drops
  The dosing regimen is every hour as needed for ear pain, not to exceed 10 mL of solution per ear in a 24-hour period
  Children 2 Months to 12 Years: dispense five drops of study drug into the affected ear canal(s) each hour, as needed for ear pain, or Children 12 years to <19 years: dispense 10 drops of study drug into the affected ear canal(s) each hour, as needed for ear pain.
  Interventions: Drug: AR01
- Glycerin ear drops (Placebo Comparator): Topical ear drops
  The dosing regimen is every hour as needed for ear pain, not to exceed 10 mL of solution per ear in a 24-hour period
  Children 2 Months to 12 Years: dispense five drops of study drug into the affected ear canal(s) each hour, as needed for ear pain, or Children 12 years to <19 years: dispense 10 drops of study drug into the affected ear canal(s) each hour, as needed for ear pain.
  Interventions: Drug: Glycerin ear drops

INTERVENTIONS:
Drug: AR01 — drops administered an needed for pain
  Other Names: benzocaine
  Arms: AR01 - Topical Otic Solution
Drug: Glycerin ear drops — placebo drops administered for ear pain
  Other Names: placebo
  Arms: Glycerin ear drops

SUMMARY:
Children ages 2 months to less than 19 years old, who have been diagnosed with a middle ear infection may receive either medicated ear drops (AR01) or glycerin (placebo) ear drops. The patient or caregiver will measure the amount of ear pain before and after the ear drops to establish if the medicated ear drops decrease the amount of pain more than the placebo ear drops. The subject may leave the clinic 60 minutes after the first dose. The ear drops can be used up to 4 days, as needed for ear pain.

DETAILED DESCRIPTION:
The study involves the initial clinic visit, using the ear drops at home and keeping a diary about the ear pain experienced and medications taken. The patient will return to the clinic 4 days later for evaluation and to return the ear drops and diary. The clinic staff will call to follow-up about the patient's condition seven days after the initial visit.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 2 mo. to < 19 yrs of age, with signs and symptoms of AOM, with moderate to severe pain (current episode 2 wks duration). Moderate to severe pain is defined as a score of 5 (on a scale of 0 - 10) on the FAECC pain scale as evaluated by a trained clinical staff or 6 (on a scale of 0 - 10) on the FPS-R as evaluated by the subject. Moderate to severe pain criteria must be met at eligibility and the pre-dose pain assessment.
* Males or non-pregnant, non-lactating females.
* The subject's caregiver must have read and signed the written informed consent (including assent from subjects 18 yrs as applicable according to Investigational review board (IRB) guidelines) prior to study participation.
* Subjects 18 yrs old must have read and signed the written informed consent prior to study participation.
* Normally active and otherwise judged to be in good health on the basis of medical history and limited physical examination.
* Females of childbearing potential must have a urine pregnancy test at the randomization visit with negative results returned prior to randomization.

Exclusion Criteria

* Perforated tympanic membrane, history of a perforated tympanic membrane in the last 6 months, or if a perforated tympanic membrane could not be ruled out by speculum examination, impedance testing tympanometry, pneumatic otoscopy, or Valsalva maneuver. Subjects who are subsequently diagnosed with a perforated membrane during treatment are to be discontinued immediately. Subjects with tympanostomy tubes are not allowed.
* Acute or chronic otitis externa.
* Chronic otitis media (refers to current episode 2 wks).
* Seborrheic dermatitis involving the affected external ear canal or pinna.
* Any otic, topical, or systemic antibiotic received within 14 days prior to study entry (topical or systemic antibiotics for acne will be allowed on a chronic basis for subjects who have been on a stable dose for at least 14 days prior to entry).
* Any topical drying agent or over-the-counter therapy for otitis media received within 36 hrs prior to enrollment.
* Known hypersensitivity to drug or similar compounds including any of the inactive ingredients.
* Subjects receiving medication on a chronic basis for pain (including steroidal or non-steroidal anti-inflammatory drugs) who have not been on a stable dose for at least 1 month prior to entry into the study.
* Clinically significant mental illness that may interfere with the conduct of the study (determined by Investigator).
* Exposure to any investigational agent within 30 days prior to study entry.
* Previous enrollment in this study.
* Subject/caregiver has a condition the Investigator believes would interfere with the ability to provide consent or assent (age-appropriate) or comply with study instructions, or that might confound the interpretation of the study results, or put the subject at undue risk.
* Subject has a glucose 6-phosphate dehydrogenase deficiency or is taking concomitant medications associated with methemoglobinemia (such as nitrates or nitrites; aniline dyes; or medications, including lidocaine, prilocaine, phenazopyridine hydrochloride [Pyridium], and others).
* Subject shows clinical signs of anemia. The absolute amount of deoxygenated or abnormal hemoglobin (rather than its percentage) is required for cyanosis to be clinically evident. Subjects with moderate-to-severe anemia may not appear cyanotic, even with elevated percentages of deoxygenated or abnormal hemoglobins.
* Subject has congenital (i.e., hereditary) methemoglobinemia.
* Subject has a recent history of acute gastroenteritis within 14 days prior to study entry.
* Subject exhibits clinical signs of methemoglobinemia, such as unexplained bluish coloring of skin, fatigue, shortness of breath, failure to thrive, and headache.
* Subjects 5 to <19 yrs old who are unable to satisfactorily complete FPS-R screening test.

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 304 (Actual)
Dates: Start 2013-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Complete ear pain relief | At or prior to 60 minutes post baseline dose
  The proportion of subjects with complete pain relief (score of 0 on Face, Activity, Ears, Cry, Consolability tool (FAECC) as measured by the Assigned Clinical Assessor or Faces Pain Scale-Revised (FPS-R) as measured by the subject prior to any analgesic/antipyretic use) at or prior to 60 minutes post baseline dose.

SECONDARY OUTCOMES:
time to complete pain relief (score of 0 on pain scales) | 10, 20, 30, 45, and a60 minutes post baseline dose
  The time to complete pain relief (score of 0 on FAECC or FPS-R prior to any analgesic/antipyretic use), in minutes.
The proportion of subjects with complete ear pain relief | at or prior to 10, 20, 30, 45, and 60 minutes post baseline dose
  The proportion of subjects with complete ear pain relief (score of 0 on FAECC or FPS-R prior to any analgesic/antipyretic use) at or prior to 10, 20, 30, 45, and 60 minutes post baseline dose.
The percent change in FPS-R and FAECC pain scores from baseline to post dose scores | measured at 10, 20, 30, 45, and 60 minutes post baseline dose
Sum of pain intensity (SPID) using FPS-R and FAECC pain scores | measured from baseline (pre-dose) to 60 minutes
Time from baseline to in-clinic use of analgesic/antipyretic to relief ear pain | 60 Minutes
The number of subjects who receive analgesic/antipyretic medications for relief of ear pain during the clinic visit | measured at or prior to 10, 20, 30, 45, and 60 minutes post baseline dose
Number of adverse events reported as a measure of safety and tolerability | up to 30 days
  measured by treatment-emergent adverse events (AEs), concomitant medications, vital signs (pulse, temperature, and respiratory rate), abbreviated physical examination (head, ears, eyes, nose and throat and chest), external ear canal and pinna for signs of local tissue toxicity, such as rash, urticaria, local burning or stinging, skin discoloration, swelling, itching, and severe redness, and an assessment for signs of methemoglobinemia (i.e., unexplained bluish coloring of skin, fatigue, shortness of breath, failure to thrive, and headache).

OTHER OUTCOMES:
Time from complete ear pain relief (score of 0 on FAECC or FPS-R) to a pain event using the home use data | up to 4 Days (± 1)
  A pain event may include analgesic/antipyretic use, a FAECC score of >/= 5 or FPS-R score of >/= 6, or study withdrawal due to AOM, treatment, or the study itself
Relation between analgesic/antipyretic use and study medication use during the in-home period | at or prior to 15, 30, and 60 minutes baseline study medication dose and up to 4 Days (± 1)
  Dates and times of analgesic/antipyretic use will be compared with the dates and times of home use of study medication to create the use or non-use outcome for each time point.

CONTACTS AND LOCATIONS:
Overall Officials: Laurence J Downey, MD, Study Chair — Arbor Pharmaceuticals, LLC
Locations (29):
- United States (29):
  - Shoals Medical Trials, Inc., Sheffield, Alabama
  - SC Clinical Research, Inc, Tuscon, Arizona
  - NEA Baptist Clinic, Jonesboro, Arkansas
  - So Cal Clinical Research Group, Bellflower, California
  - Southland Clinical Research Center, Fountain Valley, California
  - Madera Family Medical Group, Madera, California
  - Colorado Springs Health Partners /Clinical Research Advantag, Colorado Springs, Colorado
  - Pharma Research International, Inc, Naples, Florida
  - SCORE Physician Alliance, LLC, St. Petersburg, Florida
  - The Iowa Clinic, Pc, West Des Moines, Iowa
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Kentucky Pediatric / Adult Research, Bardstown, Kentucky
  - Brownsboro Park Pediatrics, Louisville, Kentucky
  - Michael W. Simon, MD, PSC, Nicholasville, Kentucky
  - Virgo-Carter Pediatrics, Silver Spring, Maryland
  - Hennepin County Medical Center -Department of Emergency Medicine, Minneapolis, Minnesota
  - Clinical Research Center, Las Vegas, Nevada
  - Valley Stream Pediatrics, Valley Stream, New York
  - White Oak Family Physicians, Asheboro, North Carolina
  - UNC Children's Hospital - General Pediatrics and Adolescent Medicine, Chapel Hill, North Carolina
  - Hometown Urgent Care and Research Center (Dayton), Dayton, Ohio
  - PMG Research of Bristol, Bristol, Tennessee
  - DiscoveResearch, Inc., Byran, Texas
  - Research Across America - Dallas, Dallas, Texas
  - Pediatric Healthcare of Northwest Houston, PA, Tomball, Texas
  - J. Lewis Research, Inc/Jordan River Family Medicine, Jordan, Utah
  - FirstMed, Salt Lake City, Utah
  - Lewis Research, Inc/Foothill Family Clinic, Salt Lake City, Utah
  - Wee Care Pediatrics, Syracuse, Utah